CLINICAL TRIAL: NCT07039435
Title: Evaluation of Frequency Allocation Tables for Recently Implanted Single-Sided Deaf Cochlear Implant Users
Brief Title: Perceptual Adaptation Following Cochlear Implantation (Aim 3a)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-01046; R01DC021980 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sensorineural Hearing Loss; Cochlear Implantation; Perceptual Adaptation
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Newly implanted Single-Sided Deaf Cochlear Implant (SSD-CI) Users (Experimental): Subjects will use four frequency maps for the first month after CI activation. One of these maps will be standard of care (i.e., 188-7938 Hz for Cochlear users) and the other three will have higher low frequency edges than the standard of care default maps (starting at 313, 438, and 563 Hz, respectively). These maps will alternate daily during the first month (with exceptions made for situations when the subject is allowed to use a preferred map rather than the map predetermined for use that day), and after that point each subject will make a selection at the beginning of the week to compare all four maps and decide which one to use at the beginning of the following week.
  Interventions: Other: Alternative Frequency Mapping

INTERVENTIONS:
Other: Alternative Frequency Mapping — Patients will have their speech processors programmed with four maps, three of which use a higher low-frequency cutoff than the default map (313 Hz, 438 Hz, 563 Hz, compared to the default map that has a low-frequency cutoff of 188 Hz).

SUMMARY:
The goal of this study is to study the adaptation process in newly implanted Single-Sided Deaf Cochlear Implant (SSD-CI) users. Subjects will use four frequency maps for the first month after CI activation. One of these maps will be standard of care and the other three will have higher low frequency edges than the standard of care default maps. These maps will alternate daily during the first month (with exceptions made for situations when the subject is allowed to use a preferred map rather than the map predetermined for use that day), and after that point each subject will make a selection at the beginning of the week to compare all four maps and decide which one to use at the beginning of the following week. The goal of this study is to investigate how reducing place-pitch mismatch in SSD CI users affects 1) sound quality, 2) device use, and 3) speech perception.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. No known anatomical abnormalities in either ear
3. English speaking
4. Intends to receive a cochlear implant in one ear (or has already received it but it has not been activated).
5. Normal hearing (or minimal hearing loss) in the contralateral ear

Exclusion Criteria:

1. Under age 18
2. Documented anatomical abnormality of the implanted ear
3. Non-English speaking
4. Greater than minimal hearing loss in the contralateral ear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Bilateral speech perception as measured by Bamford-Kowal-Bench (BKB-SIN) speech-in-noise score while using standard 188 Hz Frequency-Allocation Table (FAT) | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using standard 188 Hz FAT | 1 month post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using standard 188 Hz FAT | 3 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using standard 188 Hz FAT | 6 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using standard 188 Hz FAT | 12 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 313 Hz FAT | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 313 Hz FAT | 1 month post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 313 Hz FAT | 3 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 313 Hz FAT | 6 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 313 Hz FAT | 12 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 438 Hz FAT | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 438 Hz FAT | 1 month post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 438 Hz FAT | 3 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 438 Hz FAT | 6 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 438 Hz FAT | 12 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 563 Hz FAT | Baseline
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 563 Hz FAT | 1 month post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 563 Hz FAT | 3 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 563 Hz FAT | 6 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Bilateral speech perception as measured by BKB-SIN speech-in-noise score while using experimental 563 Hz FAT | 12 months post activation of implant
  The BKB-SIN speech-in-noise test measures speech perception in noise by assessing a listener's signal-to-noise ratio (SNR) loss. The test results are presented as the SNR loss, which is the amount the signal-to-noise ratio needs to be increased for the listener to correctly repeat 50% of the sentences. A higher SNR loss indicates more difficulty hearing.
Cochlear Implant (CI)-only speech perception as measured by the consonant-nucleus-consonant (CNC) word list score while using standard 188 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using standard 188 Hz FAT | 1 month post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using standard 188 Hz FAT | 3 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using standard 188 Hz FAT | 6 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using standard 188 Hz FAT | 12 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 313 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 313 Hz FAT | 1 month post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 313 Hz FAT | 3 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 313 Hz FAT | 6 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 313 Hz FAT | 12 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 438 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 438 Hz FAT | 1 month post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 438 Hz FAT | 3 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 438 Hz FAT | 6 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 438 Hz FAT | 12 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 563 Hz FAT | Baseline
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 563 Hz FAT | 1 month post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 563 Hz FAT | 3 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 563 Hz FAT | 6 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.
CI-only speech perception as measured by the CNC word list score while using experimental 563 Hz FAT | 12 months post activation of implant
  CNC word lists are used to evaluate the speech perception abilities of people with hearing impairments and cochlear implant users. A CNC score above 50% postoperatively indicates that a patient can communicate without relying too much on lip reading, sign language, or written communication.

SECONDARY OUTCOMES:
Sound Quality Survey score while using standard 188 Hz FAT | Baseline
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 188 Hz FAT | 1 month post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 188 Hz FAT | 3 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 188 Hz FAT | 6 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 188 Hz FAT | 12 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 313 Hz FAT | Baseline
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 313 Hz FAT | 1 month post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 313 Hz FAT | 3 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 313 Hz FAT | 6 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 313 Hz FAT | 12 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 438 Hz FAT | Baseline
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 438 Hz FAT | 1 month post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 438 Hz FAT | 3 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 438 Hz FAT | 6 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 438 Hz FAT | 12 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 563 Hz FAT | Baseline
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 563 Hz FAT | 1 month post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 563 Hz FAT | 3 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 563 Hz FAT | 6 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.
Sound Quality Survey score while using standard 563 Hz FAT | 12 months post activation of implant
  The Sound Quality Survey records subjective thoughts regarding sound quality, listening effort and intelligibility with all four maps at various time points. The survey was created for this study and consists of 4 questions address speech understanding, listening effort, sound quality, and music when the CI is ON versus when the CI is off. Items are rated from 1 (worst) to 9 (best). Scores range from 4-36, higher scores indicate better overall sound quality when the CI is on. Participants will provide a separate answers for each of the 4 maps.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A. Svirsky, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: mario.svirsky@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to mario.svirsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.